CLINICAL TRIAL: NCT06518993
Title: Observational Study to Collect Safety Data and Patient-reported Outcomes Measures (PROMs) on Retrospective Primary Total Hip Arthroplasty Surgeries With Trinity Cup and Meije Duo Cementless Hip Stem
Brief Title: Observational Study to Collect Safety Data and PROMs on Primary THA
Status: Terminated | Type: Observational
Why Stopped: The current study was prematurely terminated as part of a strategic decision to consolidate resources and incorporate the Trinity implant into another ongoing PMCF study which was initiated to meet updated regulatory requirements.
Sponsor: Corin (Industry)
Responsible Party: Sponsor
Other Study IDs: CSP2022-04
Record Dates: First submitted 2024-07-15; First posted 2024-07-25 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2025-07

CONDITIONS: Hip Arthritis; Osteoarthritis, Hip; Coxitis; Femoral Head Necrosis; Femoral Neck Fractures
Keywords: total hip arthroplasty
MeSH Terms: conditions — Osteoarthritis, Hip; Femoral Neck Fractures | interventions — Arthroplasty, Replacement, Hip

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Total hip arthroplasty with a Trinity cup and a Meije Duo cementless stem — Subjects clinically suitable for a primary THR surgery with Trinity cup and Meije Duo cementless femoral stem.

SUMMARY:
This observational study is designed to collect safety data and PROMs on retrospective primary total hipa arthroplasty surgeries with Trinity cup and Meije Duo cementless hip system

DETAILED DESCRIPTION:
The major goal of this study is to collect safety and patient-reported outcomes measures (PROMs) data on Trinity cup in combination with Meije Duo cementless hip stem when used in primary total hip arthroplasty (THA).

Data collected from this study will be fed into the Post-Market Surveillance (PMS) and Clinical Evaluation processes of the devices under assessment annually and support presentations at orthopaedic congresses and/or peer-reviewed publication(s) on mid- and long-term safety and clinical performance.

ELIGIBILITY:
Inclusion Criteria:

* Both genders.
* Adult subjects.
* Subjects who received a primary THR with Trinity cup and Meije Duo cementless femoral stem.
* The subject is willing to comply with the required follow-up visits as per protocol.
* The subject has signed a Patient Informed Consent Form (PICF), specific to this study, and approved by the local EC.

Exclusion Criteria:

* Subjects under guardianship.
* Subjects in the opinion of the Investigator/ investigative team who will be unable to comply with study procedures (Examples: recent psychotic or mania disorders, alcohol, drug or substance abusers) and/or those unable for any medical or other reason to comply with study procedures/visits.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who have undergone to a THA with Trinity cup and Meije Duo cementless hip will be invited to participate in this study. An initial review of the medical database of all Corin Trinity cup procedures performed in the selected study site will be conducted to assess the number of retrospective patients potentially available to join the study. A first contact with the patient will occur telephonically or via mail to explain the study and invite them to join.
Sampling Method: Non-Probability Sample
Enrollment: 116 (Actual)
Dates: Start 2024-04-19 (Actual); Primary Completion 2025-06-20 (Actual); Study Completion 2025-06-20 (Actual)

PRIMARY OUTCOMES:
Evaluation of hip functional performance | 2 years
  Improvement of Oxford Hip Score (OHS)

SECONDARY OUTCOMES:
Confirmation of safety of the study devices | 2 years
  Number, severity and causal relationship procedure of implant-related adverse events
Evaluation of outcome after hip arthroplasty | 2 years
  Number, severity and causal relationship procedure of implant-related adverse events
Evaluation of clinical outcomes | 2 years
  Improvement of Harris Hip Score (HHS)
Assessment of health-related quality of life | 2 years
  Change of EQ-5D-5L
Assessment of patient's satisfaction | 2 years
  Improvement of patient's satisfaction following surgery using Self-Administered Patient Satisfaction Scale

CONTACTS AND LOCATIONS:
Overall Officials: Charles BERTON, MD, Principal Investigator — CH VALENCIENNES
Locations (1):
- CH Valenciennes, Valenciennes, France

IPD SHARING:
Plan to Share IPD: No